CLINICAL TRIAL: NCT00954785
Title: The Efficacy and Safety of Administration of the COX-2 Selective NSAID, Etoricoxib (120mg od. for 7 Days) Compared to Diclofenac (50 mg Tds. for 7 Days) and Placebo as Adjunct Treatment in the First 7 Days of Treatment of Acute Grade II Lateral Ankle Ligaments Sprains: A Clinical Trial
Brief Title: Etoricoxib in Acute Ankle Ligament Sprains
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated by Merck USA. The company did not supply drugs for the study.
Sponsor: University of Cape Town (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Martin Schwellnus, Prof, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IISP 34251; Rec Ref 005/2008
Record Dates: First submitted 2009-08-06; First posted 2009-08-07 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2009-08

CONDITIONS: Sprain
Keywords: ankle; ligament; sprain; non-steroidal anti-inflammatory drugs; treatment; Acute ankle ligament sprain
MeSH Terms: conditions — Sprains and Strains | interventions — Diclofenac; tyramine-deoxysorbitol; Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo drug (Placebo Comparator)
  Interventions: Device: Ankle brace
- Etoricoxib (Experimental)
  Interventions: Device: Ankle brace; Drug: Etoricoxib 120 mg mane
- Diclofenac (Active Comparator)
  Interventions: Device: Ankle brace; Drug: Diclofenac 50 mg tds

INTERVENTIONS:
Device: Ankle brace — Sports Stirrup ankle brace (Aircast)
Drug: Diclofenac 50 mg tds — In the diclofenac group, each subject will receive 50 mg diclofenac in the morning, at mid-day and in the evening
  Other Names: Voltaren
  Arms: Diclofenac
Drug: Etoricoxib 120 mg mane — In the etoricoxib group, each subject will receive 120 mg etoricoxib in the morning, and placebo medication in the evening and at mid-day
  Other Names: Arcoxia
  Arms: Etoricoxib

SUMMARY:
The aim of the study is to measure the effectiveness of treatment over 7 days with commonly used anti-inflammatory medications namely etoricoxib and diclofenac (Voltaren) on reducing the severity of pain, swelling and loss of function (range of movement, proprioception) arising from a mild to moderate sprain (partial tear) of the lateral (outer) ligaments of the ankle joint. This injury is commonly known as an ankle sprain.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 45 years (Rationale: Most injuries occur in this age group, older subjects are more likely to have concomitant pathology e.g. osteoarthrosis)
* Acute lateral ankle ligament sprain less than 48 hours ago (Rationale: It is important to standardize the phase of the injury and enter at the time of the maximum inflammatory response, but this has to be balanced with enough time to allow injured subjects to access the treatment facility, and that all measurements can be completed)
* Grade II ankle sprain injury according to the following: (Rationale: Standard clinical criteria are used to ensure that the severity of injury is similar in all subjects)

  * Mild to moderate pain (> 40mm on the VAS)
  * Mild to moderate lateral ankle swelling (Greater than 5% increase in ankle volume compared with the uninjured side according to volumetric assessment)
  * Tenderness over the anterior talofibular ligament
* Negative urine and serum pregnancy test (females only) with signed undertaking on use of adequate contraception for the duration of the trial (Rationale: This is to make sure that no pregnant female subjects are entered or can become pregnant during the trial as a safety precaution against drug use in pregnancy)
* No use of analgesics or oral or intramuscular anti-inflammatory drugs in the last 24 hours (Rationale: This is to ensure that at the time of the first assessment, no subject has taken oral or intramuscular medication that may influence the initial assessments of pain and swelling)
* No use of topical anti-inflammatory agents, ice application or compression in the last 12 hours (Rationale: This is to ensure that at the time of the first assessment, no subject has taken topical medication, or used ice or compression that may influence the initial assessments of pain and swelling)

Exclusion Criteria:

* Patients with a history of an ankle sprain in the previous 12 months (Rationale: A recent previous injury in the ligaments may affect the healing of a new injury)
* The presence of an ankle fracture as diagnosed on normal radiographs - using the Ottowa ankle rules. (Rationale: This is to ensure that subjects only suffer from a soft tissue injury, so that the study group is homogeneous)
* Patients who have experienced bronchospasm, acute rhinitis, nasal polyps, angioneurotic oedema, urticaria, or allergic-type reactions after taking acetylsalicylic acid, NSAID's,(including COXIBS) , antipyretics or any of their excipients. (Rationale: This is to ensure that no subject who has a history of hypersensitivity to drugs is given drugs that may cause an allergic reaction)
* Patients who have a sulphonamide allergy. (Rationale: This is to ensure that no subject who has a history of hypersensitivity to certain drugs is given drugs that may cause an allergic reaction)
* Active peptic ulcer within the previous six months (Rationale: It is well established that NSAID's have gastric irritation, gastritis, and ulceration with haemorrhage as possible side effects. This is to ensure that subjects with a history of these syndromes are not included as a safety issue)
* History of recurrent peptic (gastric or duodenal) ulcer (Rationale: It is well established that NSAID's have gastric irritation, gastritis, and ulceration with haemorrhage as possible side effects. This is to ensure that subjects with a history of these syndromes are not included as a safety issue)
* History of any bleeding disorders, including gastrointestinal bleeding or cerebrovascular bleeding (Rationale: It is well established that non-selective NSAID's can decrease clotting. This is to ensure that subjects with a history of these syndromes are not included as a safety issue)
* Patients with severe congestive heart failure (NYHA 3 - 4) (Rationale: The administration of etoricoxib is contra-indicated in these patients)
* Patients with a medical history of ischemic heart disease or cerebrovascular disease. (Rationale: There is a potential risk of cardiovascular events with COX-2 selective inhibitor use, although this is only documented after long-term use (>18 months).
* History of cardiac failure, left ventricular dysfunction, hypertension or pre-existing oedema. (Rationale: Inhibition of prostaglandin synthesis, as caused by these drugs, may cause fluid retention, oedema and hypertension.
* Patients with peripheral arterial disease (Rationale: Peripheral aerial disease will alter the response to healing in the ankle ligaments)
* Patients with a history or current symptoms and clinical signs of severe impairment of renal function (CrCl <30 ml/min) or moderate to severe impairment of hepatic or function (Rationale: The administration of etoricoxib 120 mg is contra-indicated in these patients)
* Patients with inflammatory bowel disease. (Rationale: The administration of etoricoxib is contra-indicated in these patients).
* Patients consuming more than three alcoholic drinks per day, or patients with a history of alcohol abuse (Rationale: Excessive alcohol intake could negatively affect liver function, interfere with drug metabolism and reduce compliance to the protocol)
* Patients with hereditary problems of galactose intolerance, Lapp lactose deficiency or glucose-galactose malabsorption. (Rationale; etoricoxib tablets contain lactose and is therefore contraindicated in these patients)
* Currently pregnant or lactating (Rationale: The administration of etoricoxib is contra-indicated in these patients)
* Woman attempting to conceive. (Rationale: Any drug known to inhibit COX-2 is contra-indicated)
* Concomitant treatment with anti-coagulants (including heparin, warfarin, and ticlopidine) (Rationale: It is well established that NSAID's can decrease clotting. This is to ensure that subjects with a history of established bleeding disorders or those on anti-clotting therapy are not included as a safety issue).
* Concomitant treatment with lithium, methotrexate, angiotensin converting enzyme inhibitors, beta-blockers and diuretics) (Rationale: NSAID's have significant drug interactions with some medications, can potentiate or impair the effects of others and therefore patients on these medications are excluded for safety reasons).
* Concomitant administration of other NSAID's (including aspirin doses > 150 mg) or analgesic agents (Rationale: The purpose of the study is to determine the effects of specific NSAID's on pain and swelling. Concomitant use of other NSAID's will interfere with outcome measures and these patients have to be excluded from the study)
* Concomitant administration of cyclosporine and tacrolimus. (Rationale: Co-administration of these medications with any NSAID's may increase their nephrotoxic effects)
* Concomitant treatment of etoricoxib with rifampicin. (Rationale: Rifampicin is a potent inducer of CYP enzymes and produces a 65% decrease in etoricoxib plasma concentration.)
* Current treatment or treatment within the last two months with corticosteroids (systemic, intra-articular) (Rationale: Long acting corticosteroids can interfere with outcome measures and patients who received these medications have to be excluded from the study)
* Participation in another clinical trial during this study or during the previous month (Rationale: This is to ensure that patients who may still have effects from treatment administered during another trial are not included)
* Inability to comply with the protocol (Rationale: This is to exclude subjects who will not be able to complete the study)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Pain | 7 days

SECONDARY OUTCOMES:
Swelling | 7 days
Range of motion | 7 days
Proprioception | 7 days
Adverse events | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Martin P Schwellnus, MBBCh, MD, Principal Investigator — University of Cape Town
Locations (2):
- South Africa (2):
  - Kuilsriver Netcare Hospital, 33 Van Riebeeck Road, Kuilsriver, Cape Town, Western Cape
  - Sports Medicine Clinic, Sports Science Institute of South Africa, Cape Town, Western Cape

REFERENCES:
- [Derived] Jones P, Lamdin R, Dalziel SR. Oral non-steroidal anti-inflammatory drugs versus other oral analgesic agents for acute soft tissue injury. Cochrane Database Syst Rev. 2020 Aug 12;8(8):CD007789. doi: 10.1002/14651858.CD007789.pub3. PMID 32797734